CLINICAL TRIAL: NCT05345522
Title: A Single-arm, Open-label, Multi-center Phase Ⅱa Clinical Study to Evaluate the Efficacy and Safety of Recombinant Humanized Anti-IL-6R mAb Injection in the Treatment of Patients With Idiopathic Multicentric Castleman's Disease
Brief Title: A Study of Anti-IL-6R mAb Injection in Patients With iMCD
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Beijing VDJBio Co., LTD. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: VDJ001-MCD-Ⅱa
Record Dates: First submitted 2022-04-19; First posted 2022-04-26 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Idiopathic Multicentric Castleman's Disease
Keywords: anti IL-6R; iMCD

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- Recombinant Humanized Anti-interleukin-6 Receptor Monoclonal Antibody Injection 4 mg/kg, q2w (Experimental): Recombinant Humanized Anti-interleukin-6 Receptor Monoclonal Antibody Injection 4 mg/kg as the low dose group in phase I.
  Interventions: Biological: Recombinant Humanized Anti-interleukin-6 Receptor Monoclonal Antibody Injection 4 mg/kg, q2w
- Recombinant Humanized Anti-interleukin-6 Receptor Monoclonal Antibody Injection 6 mg/kg, q2w (Experimental): Recombinant Humanized Anti-interleukin-6 Receptor Monoclonal Antibody Injection 6 mg/kg, q2w as the middle dose group in phase I.
  Interventions: Biological: Recombinant Humanized Anti-interleukin-6 Receptor Monoclonal Antibody Injection 6 mg/kg, q2w
- Recombinant Humanized Anti-interleukin-6 Receptor Monoclonal Antibody Injection 8 mg/kg, q2w (Experimental): Recombinant Humanized Anti-interleukin-6 Receptor Monoclonal Antibody Injection 8 mg/kg, q2w, as the high dose group in phase I.
  Interventions: Biological: Recombinant Humanized Anti-interleukin-6 Receptor Monoclonal Antibody Injection 8 mg/kg, q2w
- Recombinant Humanized Anti-interleukin-6 Receptor Monoclonal Antibody Injection 6 mg/kg, q3w (Experimental): Recombinant Humanized Anti-interleukin-6 Receptor Monoclonal Antibody Injection 6 mg/kg, q3w, as the high dose group in phase II.
  Interventions: Biological: Recombinant Humanized Anti-interleukin-6 Receptor Monoclonal Antibody Injection 6 mg/kg, q3w
- Recombinant Humanized Anti-interleukin-6 Receptor Monoclonal Antibody Injection 4mg/kg, q3w (Experimental): Recombinant Humanized Anti-interleukin-6 Receptor Monoclonal Antibody Injection 4mg/kg, q3w, as the low dose group in Phase II.
  Interventions: Biological: Recombinant Humanized Anti-interleukin-6 Receptor Monoclonal Antibody Injection 4mg/kg,q3w

INTERVENTIONS:
Biological: Recombinant Humanized Anti-interleukin-6 Receptor Monoclonal Antibody Injection 4 mg/kg, q2w — Recombinant Humanized Anti-interleukin-6 Receptor Monoclonal Antibody Injection 4 mg/kg, intravenous injection for 60 to 90 minutes. Every 2 weeks is a cycle, the first day of each cycle is administered, a total of ≥ 4 cycles.
  Arms: Recombinant Humanized Anti-interleukin-6 Receptor Monoclonal Antibody Injection 4 mg/kg, q2w
Biological: Recombinant Humanized Anti-interleukin-6 Receptor Monoclonal Antibody Injection 6 mg/kg, q2w — Recombinant Humanized Anti-interleukin-6 Receptor Monoclonal Antibody Injection 6 mg/kg, intravenous injection for 60 to 90 minutes. Every 2 weeks is a cycle, the first day of each cycle is administered, a total of ≥ 4 cycles.
  Arms: Recombinant Humanized Anti-interleukin-6 Receptor Monoclonal Antibody Injection 6 mg/kg, q2w
Biological: Recombinant Humanized Anti-interleukin-6 Receptor Monoclonal Antibody Injection 8 mg/kg, q2w — Recombinant Humanized Anti-interleukin-6 Receptor Monoclonal Antibody Injection 8 mg/kg, intravenous injection for 60 to 90 minutes. Every 2 weeks is a cycle, the first day of each cycle is administered, a total of ≥ 4 cycles.
  Arms: Recombinant Humanized Anti-interleukin-6 Receptor Monoclonal Antibody Injection 8 mg/kg, q2w
Biological: Recombinant Humanized Anti-interleukin-6 Receptor Monoclonal Antibody Injection 4mg/kg,q3w — Recombinant Humanized Anti-interleukin-6 Receptor Monoclonal Antibody Injection 4 mg/kg, intravenous injection for 60 to 90 minutes. Every 3 weeks is a cycle, the first day of each cycle is administered, a total of ≥ 4 cycles.
  Arms: Recombinant Humanized Anti-interleukin-6 Receptor Monoclonal Antibody Injection 4mg/kg, q3w
Biological: Recombinant Humanized Anti-interleukin-6 Receptor Monoclonal Antibody Injection 6 mg/kg, q3w — Recombinant Humanized Anti-interleukin-6 Receptor Monoclonal Antibody Injection 6 mg/kg, intravenous injection for 60 to 90 minutes. Every 3 weeks is a cycle, the first day of each cycle is administered, a total of ≥ 4 cycles.
  Arms: Recombinant Humanized Anti-interleukin-6 Receptor Monoclonal Antibody Injection 6 mg/kg, q3w

SUMMARY:
This study is a single-arm, open-label, multicenter, dose-escalation clinical study. Its primary purpose is to evaluate the safety and tolerability of recombinant humanized anti-interleukin-6 receptor monoclonal antibody ( Anti-IL-6R mAb ) injection in patients with Idiopathic Multicentric Castleman's Disease ( iMCD ) and to determine the recommended dose for follow-up studies. Its secondary purpose is to evaluate the preliminary efficacy, immunogenicity and pharmacokinetic ( PK ) index, pharmacodynamic ( PD ) characteristics of Anti-IL-6R mAb injection in patients with iMCD.

DETAILED DESCRIPTION:
Phase I:

This stage is a single-arm, open-label, multicenter, dose-escalation clinical study. A total of 3 dose groups of 4 mg/kg, 6 mg/kg and 8 mg/kg, 3 patients per dose, are designed in this study to explore the safety, tolerability and preliminary efficacy of the experimental drug administered for ≥4 cycles in patients with iMCD. Referring to the inclusion and exclusion criteria, the patients will be enrolled from the low-dose group to the high-dose group in turn. After the last patient of each dose group completed the third administration and 2-week safety observation, the investigator and the sponsor will discuss the safety results of the patients together in this dose group. If no any important adverse event occurs, they can enter the next dose group. If an important adverse event occurs in any patient, the investigator and the sponsor will discuss whether to continue the study in the next dose group. Dose escalation will be discontinued if more than one patient experiences an important adverse event. If an important adverse event occurs, the investigator will perform related inspections based on the patient's condition, and for treatment.

After the patient completes four cycles of administration, if no significant safety events are found or the patient has not withdrawn from the trial due to significant safety events and has a significant treatment effect, and if the investigator determines that they may benefit from continuing the treatment, with the consent of both the investigator and the patient.

Phase I is planned to include 9 patients.

Phase II:

This stage is a single-arm, open-label, multicenter clinical study. Based on the analysis of all patients' data up to C10D14 from the first stage, it is planned to further explore the dosing regimens of 4 mg/kg and 6 mg/kg in this stage. A total of two groups are set up. Group 1: 4 mg/kg, 1 cycle every 3 weeks, 1 dose per cycle, administered on the first day of each cycle, if the investigator assesses that the poor efficacy may be caused by insufficient dose, after communication with the sponsor, the patient can be transferred to the 6 mg/kg dose group for continued treatment observation to explore the safety and preliminary efficacy of the investigational drug when administered for ≥ 4 cycles in iMCD patients; Group 2: 6 mg/kg, 1 cycle every 3 weeks, 1 dose per cycle, administered on the first day of each cycle, to explore the safety and preliminary efficacy of the investigational drug when administered for ≥ 4 cycles in iMCD patients. According to the inclusion and exclusion criteria, 8 patients were enrolled in each group 1 and group 2. Patients were enrolled in sequence according to the number, and the first 8 patients were enrolled in group 1, and the next 8 patients were enrolled in group 2.

After 4 cycles of administration in patients of group 1 or group 2, if the treatment effect is obvious and the investigator judges that the patient may benefit from continuing the treatment, with the consent of both the investigator and the patient, the patient enters the extension period.

Phase II is planned to include 16 patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old, gender is not limited;
2. Biopsy or center pathology examination confirmed the measurable, symptomatic iMCD (iMCD diagnosis based on The consensus of the diagnosis and treatment of Castleman disease in China (2021));
3. Clinical laboratory test values within 4 weeks before treatment meet the following criteria:

   Absolute neutrophil count (ANC)≥1.0×10^9/L; Platelet count (Plt) ≥ 75×10^9/L; Alanine aminotransferase (ALT) < 2.5×upper limit of normal (ULN) ; Total bilirubin (TBIL) <2.5×ULN; Serum creatinine (Scr) ≤ 3.0 mg/dL (265 umol/L).
4. ECOG-PS physical status score of 0, 1 or 2 points;
5. When using corticosteroids, the dose of prednisone should not exceed 1 mg/kg/day (or equivalent dose), and the dose should be maintained or reduced within 4 weeks before the first dose;
6. Patients of childbearing age (males and females) must agree to take effective contraceptive measures during the trial and within 3 months after the last medication, males are not allowed to donate sperm, and females are not allowed to donate eggs;
7. The patients themselves (or their legally recognized representatives) must sign an informed consent form before performing any research-specific procedures, indicating that they understand the purpose of the research and the procedures that need to be performed, and voluntarily participate in this research.

Exclusion Criteria:

1. Human immunodeficiency virus (HIV) or human herpesvirus 8 (HHV-8) positive;
2. Skin lesions are the only detectable lesions;
3. Patients with concurrent malignant tumors (disease-free time < 5 years), except for the following cases: fully treated skin basal cell carcinoma or squamous cell carcinoma, cervical carcinoma in situ;
4. Patients with diseases that may interfere with the research process or research results, such as autoimmune diseases (systemic lupus erythematosus, rheumatoid arthritis, adult Still's disease, juvenile idiopathic arthritis, autoimmune lymphoproliferative syndrome) ), active systemic infection, poorly controlled diabetes, acute diffuse infiltrative lung disease;
5. Those who use contraindicated treatments or plan to use the following treatments during the study period:

   Received IL-6 or IL-6R targeted drug therapy before the first dose; Received other concomitant anti-tumor therapy for Castleman's disease (such as anti-CD20 antibody, chemotherapy) within 8 weeks before the first dose; Received biologics such as anti-tumor necrosis factor-α (TNF-α) antibodies within 8 weeks before the first dose; Received immunosuppressive agents (other than stable doses of corticosteroids) within 8 weeks prior to the first dose; Received erythropoiesis-stimulating agents (ESAs) within 8 weeks prior to the first dose; Received any systemic therapy for Castleman's disease within 4 weeks prior to the first dose; Major surgery or radiotherapy within 4 weeks before the first dose; Are receiving or planning to receive treatment with a strong CYP3A inhibitor during the study period.
6. Uncontrolled history of heart disease, such as unstable angina, congestive heart failure, myocardial infarction within the past 12 months, hemodynamic instability or known left ventricular ejection fraction (LVEF) <40% or clinically significant cardiac rhythm or conduction abnormalities;
7. Persons with positive infectious disease test (positive hepatitis B surface antigen (HBsAg) and hepatitis B virus-DNA titer>1000IU/ml, hepatitis C virus , syphilis, active pulmonary tuberculosis);
8. History of allogeneic transplantation (except corneal transplantation);
9. Those who are known to have severe infusion reactions to monoclonal antibodies or murine, chimeric or human proteins;
10. Pregnant or lactating women, or those who plan to become pregnant within 3 months after the last dose;
11. Those who have been vaccinated with the new coronavirus vaccine or other live attenuated vaccines within 4 weeks before the first administration, or who plan to be vaccinated during the trial period;
12. Those who have participated in other clinical trials within 1 month before the first administration;
13. Patients with paraneoplastic pemphigus or bronchiolitis obliterans;
14. Patients with a history of bleeding，including:

    Intracranial hemorrhage within 6 months before screening; Active bleeding within 2 months prior to screening.
15. Patients with cerebral infarction within 6 months before screening (except lacunar infarction);
16. Any other circumstances judged by the investigator to be inappropriate to participate in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2022-04-18 (Actual); Primary Completion 2022-11-27 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events(AEs) as Assessed by CTCAE v5.0 | Through study completion, an average of 3 years in Phase I and 1 year in phase II
  An AE is any untoward medical occurrence in a clinical study participant administered a medicinal product. The AE can be any symptom, disease or abnormal laboratory finding, which does not necessarily have a causal relationship with this treatment.
Grades of all the Adverse Events(AEs) by CTCAE v5.0 | Through study completion, an average of 3 years in Phase I and 1 year in phase II
  Grade refers to the severity of the AE. The CTCAE displays Grades 1 through 5 with unique clinical descriptions of severity for each AE based on this general guideline.

SECONDARY OUTCOMES:
Percentage of Participants Who Achieved Overall Response Rate（ORR）for Biochemical Response | Through study completion, an average of 3 years in Phase I and 1 year in phase II
  ORR is CR + PR. Biochemical indicators include 4 laboratory test indicators, namely C-reactive protein, hemoglobin, albumin and glomerular filtration rate. CR is the return of 4 biochemical indicators to normal. PR is a greater than 50% improvement in all four biochemical parameters.
Percentage of Participants Who Achieved Overall Response Rate（ORR）for Lymph Nodes | Through study completion, an average of 3 years in Phase I and 1 year in phase II
  ORR is Complete Response (CR) + Partial Response (PR) , assessed according to International Working Group ( IWG ) 1999 criteria.
Percentage of Participants Who Achieved Overall Response Rate（ORR）for Symptomatic Response | Through study completion, an average of 3 years in Phase I and 1 year in phase II
  ORR is CR + PR. The symptom response involves 4 symptoms, namely fatigue, anorexia, fever, and weight loss. CR is 4 symptoms returning to pre-onset. PR is improvement in all 4 symptoms, but not return to pre-onset.
Concentration of Anti-Drug Antibody (ADA) | Through study completion, an average of 2 years in Phase I and 1 year in phase II
  The concentrations of ADA in serum will be tested.
Concentration of Neutralizing Antibody (NAb) | Through study completion, an average of 2 years in Phase I and 1 year in phase II
  The concentration of NAb in serum will be tested when their ADA is positive.
Concentration of Soluble Interleukin-6 Receptor (sIL-6R) | Through study completion, an average of 2 years in Phase I and 1 year in phase II
  The concentrations of sIL-6R in the serum of each subject are measured.
Concentration of Interleukin-6 (IL-6) | Through study completion, an average of 2 years in Phase I and 1 year in phase II
  The concentrations of IL-6 in the serum of each subject are measured.
Cmax | Through study completion, an average of 2 years in Phase I and 1 year in phase II
  Peak concentration. Obtain directly according to the measured data of blood concentration-time.
AUC0-t | Through study completion, an average of 2 years in Phase I and 1 year in phase II
  The area under the curve from time zero to the last time that the blood drug concentration can be quantitatively detected.

CONTACTS AND LOCATIONS:
Overall Officials: Jian li, M.D., Principal Investigator — Peking Union Medical College Hospital
Locations (3):
- China (3):
  - Peking Union Medical College Hospital, Beijing
  - Peking University First Hospital, Beijing
  - West China Hospital of Sichuan Hospital, Chengdu

IPD SHARING:
Plan to Share IPD: No